CLINICAL TRIAL: NCT03866889
Title: Efficacy of an Intervention Through a Guided Training Program of Maximum Strength, in the Improvement of the Functionality of the Lower Member in Military Personnel. A Randomized Clinical Trial
Brief Title: Guided Training Program of Maximum Strength in Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SOLDUNI project
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Military Activity
Keywords: Strength; Military; Functionality; Physiotherapy; Randomized clinical trial
MeSH Terms: interventions — pamabrom

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength (Experimental): Maximum strength protocol based on a Maximum Repetition (1RM). The aim of the application of the training is to produce an increase in strength based on training with high loads (80% 1RM), individually and covering the muscles of the lower extremity (quadriceps, hamstrings, gluteus maximus).
  Interventions: Other: Strength
- Normal activity (Active Comparator): The subjects included in the control group will perform the same physical activity to improve the strenght until the beginning of the study. The exercises will be done in the same conditions and with the same period (4 days / week)
  Interventions: Other: Normal activity

INTERVENTIONS:
Other: Strength — In the performance of the squat exercise (Back Squat), the subjects will be standing, with an Olympic bar behind their neck, supported on both trapezoids, while the hands will help to hold and stabilize the bar, taking it from below.
  For hamstring curl, the subject will be in the prone position, clinging to the backrest, with the legs under the arm that lifts the weight.
  The deadlift exercise will be performed from the standing posture, holding the bar with your arms extended and the trunk straight, while your hands will hold the bar at the height and separation of the hips.
  Finally, in the quadriceps chair the subject will find himself sitting with his back straight and supported on the back of the seat, while the legs will go under the arm that lifts the weight.
  Other Names: Maximum strength
  Arms: Strength
Other: Normal activity — The subjects included in the control group will continue to perform the same strength training plan that they did before starting this one. The periodicity will be the same (4 days / week) and with the same intensity.
  Other Names: Maximum strength
  Arms: Normal activity

SUMMARY:
Introduction. The members of the Military Emergency Unit must be physically prepared for any type of situation where required, although their strength training does not follow any concrete structure. Structured training of maximum strength aims to increase the recruitment of different types of fibers, and the increase in the size of these.

Objectives: To evaluate the effectiveness of a maximum strength training protocol in lower extremity functionality in military personnel aged 25 to 45 years.

Study design. Randomized, single-blind clinical study with follow-up period. Methodology. 65 male subjects will be recruited, who will be randomly assigned to the two study groups: experimental (structured strength training) and control (they will continue with their usual routine of free training). The intervention will last for 8 weeks, with 2 weekly sessions, lasting 20 minutes, with three evaluations (baseline, posttreatment and follow-up). The study variables will be: lower limb functionality (assessed by Standing Long Jump and Single Leg Hop tests), and quadriceps and hamstring strength (evaluated with the MRI measurement for each exercise). To perform the analysis of normality, the Kolmogorov Smirnof test will be used. In case of homogeneity, with the t-student test of repeated measures and an ANOVA of repeated means, the difference between the different evaluations and the intra and intersubject effect, respectively, will be calculated.

Expected results. Effectiveness of structured training of maximum strength in functionality of lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* Military personnel belonging to the Military Emergency Unit
* male
* With an age of 25 to 45 years
* No history of musculoskeletal injury in the 3 months prior to the study

Exclusion Criteria:

* Present a diagnosis of injury in the period prior to or during the study
* Who are receiving a physiotherapy intervention at the time of the study
* Not signed the informed consent document

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Maximum strength after treatment and at one month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The RM strength assessment protocol will be used. In the squat you will be asked to bend your knees and hips over ninety degrees, then return to the starting position. In deadlift, you will be asked to take the bar from the height of the hips to just below the label, keeping the trunk upright, facing the front. Both in the quadriceps chair and in the hamstring curl, you will be asked to perform the lifting of the indicated weight, following the movement allowed by the machine to be used. The greater the weight lifted (in kg), the greater muscular strength.

SECONDARY OUTCOMES:
Change from baseline lower limb functionality after treatment and at one month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the lower limb functionality will be carried out by Standing Long Jump.In the use of Standing Long Jump, with the subject standing, behind a demarcated line aligns the tips of the feet, a squat will be requested by throwing the arms backwards and ordering the performance of a bipodal jump, with impulse of the extremities inferior ones, helping themselves with the balancing of the superiors. The distance traveled will be measured in centimeters and the test will only be valid when the subject lands with both limbs without losing balance. At greater distance (cm), greater functionality of lower limbs.
Change from baseline lower limb functionality after treatment and at one month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The functionality was measured with the Standing Long Jump test, with the subject standing, behind a demarcated line aligns the tips of the feet. You will be asked to squat by throwing your arms behind you and ordering a bipodal jump, with impulse of the lower limbs being helped by the swing of the upper ones. The distance traveled will be measured in centimeters and the test will only be valid when the subject lands with both limbs without losing balance. The measurement is made from the starting line to the landing point coinciding with the tip of the subject's feet. This test is done in a monopodal way. At greater distance (cm), greater functionality of lower limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain